CLINICAL TRIAL: NCT04577989
Title: Clinical Comparison of Treatment Strategies in AmpC Beta-lactamase Producing Enterobacterales in a Swiss Tertiary Care Hospital (AmpC-strat Basel)
Brief Title: Clinical Comparison of Treatment Strategies in AmpC Beta-lactamase Producing Enterobacterales in a Swiss Tertiary Care Hospital
Acronym: AmpCstratBasel
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02251; me20TschudinSutter
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Infection With AmpC Beta-lactamase Producing Enterobacterales
Keywords: antibiotic resistance; Ambler class C beta-lactamase (AmpC); carbapenem resistance; minimum inhibitory concentrations (MICs); cefepime; piperacillin/tazobactam; carbapenem; Clostridium difficile infections; epidemiological trends
MeSH Terms: conditions — Clostridium Infections | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection — data collection for treatment strategies (cefepime vs. piperacillin/tazobactam vs. carbapenems) of infections caused by AmpC beta-lactamase producing Enterobacterales for the period January 1st , 2015 until July 31st , 2020.

SUMMARY:
This study is to investigate the recent epidemiological trends and the treatment outcome in terms of the length of hospital stay, the relevant renal and neurological side effects, risk factors for developing these side effects, the selection of more resistant pathogens under therapy as well as the incidence of Clostridium difficile infections under treatment.

DETAILED DESCRIPTION:
Increasing resistance among Enterobacterales to beta-lactam antibiotics is globally a major concern in the antibiotic resistance crisis. In gram-negative bacteria it evolves primarily through the production of beta-lactamases that allow the rapid hydrolysis of common antibiotics - most notably 3rd generation cephalosporins. Particularly, the production of Ambler class C beta-lactamase (AmpC) is a very concerning and unique resistance mechanism as so called derepressed mutants can be induced during treatment. Information on recent epidemiological trends as well as comparative information about the treatment strategies (cefepime versus piperacillin/tazobactam versus carbapenems) for infections with AmpC-producing Enterobacterales in Switzerland is still lacking. This study is to investigate the recent epidemiological trends and the treatment outcome in terms of the length of hospital stay, the relevant renal and neurological side effects, risk factors for developing these side effects, the selection of more resistant pathogens under therapy as well as the incidence of Clostridium difficile infections under treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with detection of AmpC beta-lactamase producing Enterobacterales

  1. In a blood culture (any ward)
  2. In a clinical sample of the lower respiratory tract (only intensive care unit)

Exclusion Criteria:

* Patients with documented refusal of subsequent use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the inpatient setting at the University Hospital Basel from January 1st, 2015 until July 31st, 2020 with detection of AmpC beta-lactamase producing Enterobacterales
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
descriptive analyses of demographic data in patients with detection of AmpC beta-lactamase producing Enterobacterales | single time-point at baseline
  collection of demographic data (age, gender, hospital admission and discharge date, length of stay, ICU-stay, hospitalization prior to current hospital stay, discharge destination, outcome, cause of death, travel); descriptive analyses summarized as counts
descriptive analyses of clinical data in patients with detection of AmpC beta-lactamase producing Enterobacterales | single time-point at baseline
  descriptive analyses of clinical data (comorbidities, renal function, previous exposure to antibiotics and proton pump inhibitors, immunosuppressive treatment, date of diagnosis and type of infection with AmpC producing Enterobacterales) summarized as counts
descriptive analyses of treatment data in patients with detection of AmpC beta-lactamase producing Enterobacterales | single time-point at baseline
  descriptive and comparative analyses of treatment data (empiric and definitive antibiotic therapy including dosage, date of initiation/ discontinuation and changes in antibiotic therapy, exposures to other antimicrobials, concomitant medication, side effects) summarized as counts
descriptive analyses of microbiological data in patients with detection of AmpC beta-lactamase producing Enterobacterales | single time-point at baseline
  descriptive analyses of microbiological data Species of AmpC producing Enterobacterales, type of sample, date of sample, history of colonization or infection with any antibiotic resistant pathogen, Gram-staining of endotracheal aspirate or bronchoalveolar lavage (BAL), neutrophile and epitheliale cell count, results of culture from sputum, endotracheal aspirate, BAL or lung tissue) summarized as counts

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tschudin Sutter, Prof. Dr. med., Principal Investigator — Division of Infectious Disease and Hospital Epidemiology,University Hospital Basel
Locations (1):
- Division of Infectious Disease and Hospital Epidemiology, University Hospital Basel, Basel, Switzerland